CLINICAL TRIAL: NCT06413238
Title: Investigating the Effects of Curcumin and Saffron on Fertility, Sugar, Lipid and Anthropometric Indicators in Women With Diabetes Mellitus of Reproductive Age
Brief Title: Rationale and Design of Diabetes Management With Curcumin and Saffron (DMCS): a Randomised, Three Blind -Blind, Placebo-controlled Study
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fateme Moshirenia (Other)
Collaborators: Tarbiat Modarres University (Other)
Responsible Party: Sponsor-Investigator, Fateme Moshirenia, Department of Midwifery & Reproductive Health, Medical Sciences Faculty, Tarbiat Modares University, Tehran, Iran, Tarbiat Modarres University
Organization: Tarbiat Modarres University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: fatememoshirenia4420185791; f.moshirenia40120262004 (Registry Identifier: curcuminsaffaron)
Record Dates: First submitted 2024-05-05; First posted 2024-05-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Women of Reproductive Age; Diabetes Mellitus
Keywords: diabetes; reproductive age; curcumin; saffron; lipid profile; sugar profile; enterometric indices
MeSH Terms: conditions — Diabetes Mellitus | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: In Arm curcumin, participants will receive two curcumin capsules, each with a dose of 500 mg, in addition to routine treatments. In Arm saffaron, participants will use one 15 mg saffron capsule and one placebo capsule, in addition to routine treatments. In Arm combination, participants will use one 500 mg curcumin capsule and one 15 mg saffron capsule, in addition to routine treatments. In Arm plasebo , participants will use two placebo capsules (500 mg starch flour), in addition to routine treatments
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will involve capsules with different combinations of curcumin, saffron, and placebos, labeled as ABCD. The capsules will be identical in appearance and smell to maintain blinding. The researcher, participants, and pharmacist will be unaware of the capsule contents. This three-way blind method aims to eliminate bias in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- curcumin (Other): curcumin
  Interventions: Drug: curcumin, saffron, Combination of saffron and curcumin and placebo
- saffron (Other): saffron
  Interventions: Drug: curcumin, saffron, Combination of saffron and curcumin and placebo
- Combination (Other): Combination of saffron and curcumin
  Interventions: Drug: curcumin, saffron, Combination of saffron and curcumin and placebo
- placebo (Placebo Comparator): placebo
  Interventions: Drug: curcumin, saffron, Combination of saffron and curcumin and placebo

INTERVENTIONS:
Drug: curcumin, saffron, Combination of saffron and curcumin and placebo — This study investigates the individual and combined effects of curcumin and saffron on diabetes compared to a placebo group. It will assess the effects on both clinical and laboratory diabetes symptoms within and between groups. Participants will receive either two 500mg curcumin capsules in arm 1, one 15mg saffron capsule with a 500mg starch flour placebo in arm 2, one 500mg curcumin and one 15mg saffron capsule in arm 3, and two 500mg starch flour placebos in arm 4.

SUMMARY:
## Study Hypotheses Summary:

**Primary Hypothesis:** Women with diabetes mellitus receiving the intervention will exhibit significantly lower levels of sugar indicators (FBS, HA1c, 2HPP) and lipid indicators (LDL, HDL, TG) compared to the placebo group.

**Secondary Hypotheses:**

1. **Psychological Outcomes:** The intervention group will show significant reductions in stress, anxiety, and depression compared to the placebo group.
2. **Sexual Health Outcomes:** The intervention group will experience improvements in sexual performance, marital satisfaction, and quality of sexual life compared to the placebo group.
3. **Diabetes Management Outcomes:** The intervention group will demonstrate improvements in clinical symptoms of diabetes and anthropometric index compared to the placebo group.
4. **Medication Adherence:** The intervention will be well-received by women with diabetes mellitus of reproductive age, leading to improved medication adherence.

DETAILED DESCRIPTION:
The study is a four-arm trial testing the effectiveness of curcumin, saffron, and a combination of both compared to a placebo in women with diabetes. The trial will measure glucose and lipid levels, medication side effects, adherence to treatment, and various other health indicators at different time points. Participants will be recruited from a specialty diabetes clinic in Yazd province, Iran, with specific eligibility criteria including age, diabetes diagnosis, and exclusion criteria such as allergies and certain medication use. The diagnostic criteria for diabetes mellitus are outlined by the American Diabetes Association.

ELIGIBILITY:
Inclusion Criteria:

* being married, having type 2 diabetes(according to American Diabetes Association provides guidelines) that had been diagnosed and treated for at least one year, not being dependent on insulin, being between the ages of 18-45 and having a body mass index between 18.5 and 30. Additionally, Absence of menorrhagia on the basis of the PBLAC chart

Exclusion Criteria:

* Participants who are allergic to turmeric or saffron plant essence will be excluded from the study. Additionally, women who do not regularly use supplements or take drugs for at least 7 consecutive days per month were excluded. Anticoagulant use, pregnancy, and breastfeeding will be also exclusion criteria. Finally, participants who had taken multivitamins or supplements affecting metabolism in the last three months will be not included in the study. Exclusion criteria for the study will include changes in diet and physical activity, experiencing a stressful event during the intervention (as reported by the research unit), and the use of drugs that affect sexual performance (as reported by the research unit)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with diabetes mellitus of reproductive age
Enrollment: 120 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-22 (Estimated)

PRIMARY OUTCOMES:
Sugar and lipid indicators | Sugar and lipid indicators will be measured at baseline Post-intervention .
  Sugar and lipid indicators will be measured using Delta DP diagnostic kits. The Delta DP diagnostic kits have an inter-assay CV of <3% and an intra-assay CV of <2%, indicating highly accurate and reliable test results within the same assay and between different assays.

SECONDARY OUTCOMES:
stress, anxiety and depression | at baseline ,Completion of the intervention and Follow up period (6 weeks after Completion of the intervention)
  stress, anxiety, and depression will be measured by DASS21 questionnaire
Sexual performance | at baseline ,Completion of the intervention and Follow up period (6 weeks after Completion of the intervention)
  Sexual performance will be FSFI questionnaire
quality of sexual | at baseline ,Completion of the intervention and Follow up period (6 weeks after Completion of the intervention)
  quality of sexual life will be measured by SQOL-F questionnaire
marital satisfaction | at baseline ,Completion of the intervention and Follow up period (6 weeks after Completion of the intervention)
  marital satisfaction will be measured by SQOL-F questionnaire
adherence to treatment | at baseline ,Completion of the intervention and Follow up period (6 weeks after Completion of the intervention)
  adherence to treatment will be measured by Morisky questionnaire

IPD SHARING:
Plan to Share IPD: Yes
starting 6 months after publication
Supporting Information: Study Protocol, ICF